CLINICAL TRIAL: NCT00600392
Title: Transcriptomal Analysis of Peripheral Blood and Skeletal Muscle in Patients Undergoing CRT Using Oligonucleotide Arrays
Brief Title: DNA/RNA Analysis of Blood and Skeletal Muscle in Patients Undergoing Cardiac Resynchronization Therapy (CRT)
Acronym: Medusa PH
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00009277; 7523 (Other: Duke legacy protocol number)
Record Dates: First submitted 2008-01-15; First posted 2008-01-25 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2012-11

CONDITIONS: Cardiomyopathy (Ischemic or Non-Ischemic)
MeSH Terms: conditions — Cardiomyopathies; Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum TNF alpha, IL-1, IL6, CRP, uric acid, albumin, BNP, IGF-1 and growth hormone at baseline and at 6 months.
  50 ml of blood will be collected at baseline and at 6 months. It will be divided into aliquots as follows; 10 ml in Pax-gene tubes for mRNA extraction, 20 ml for various other biomarkers, 10 ml for proteomics and 10 ml will be stored for any future use.
  Approximately a 5x5 - 7x7mm muscle biopsy will be obtained from the mid thigh region of each subject at baseline and at six months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: patients who meet criteria for CRT-D implantation

SUMMARY:
Genes expressing inflammatory cytokines (TNF- alpha, IL1 etc) and genes involved in apoptosis (Caspase 3, Bax, Bcl-2, Fas) are dysregulated in the skeletal muscles of the patients who have muscle wasting and decreased exercise capacity with CHF.

Patients who show benefit from CRT may also show reversal of the inflammatory/apoptotic cascade that accompanies CHF and these patients may be the ones who benefit the most from CRT

DETAILED DESCRIPTION:
1. The general objective of this study is to:

1. To identify the molecular pathways that may be altered in the blood and skeletal muscles of the patients undergoing CRT by using transcriptional analysis of the blood and skeletal muscle in these patients
2. To identify objective measurable molecular signals, using gene expression profiling, that correlate with clinical improvement in patients undergoing CRT.
3. To identify the molecular profile of patients who are most likely to benefit from CRT with improvement of exercise capacity and reversal of cardiac cachexia.
4. To identify biochemical pathways involved in cardiac cachexia.
5. To identify genes involved in positive remodeling and reversal of apoptotic cascade in the skeletal muscle.

ELIGIBILITY:
Inclusion Criteria:

* Patients with poor LV function and an EF of ≤35%
* Patients who are symptomatic with Class II or Class III heart failure on optimal medical therapy.
* Patients with EKG showing QRS duration of greater than 120 ms and meet criteria for Bi-ventricular ICD implantation.

Exclusion Criteria:

* Patients with other co-morbid conditions which could contribute to cachexia, such as end stage renal disease, ongoing malignancy, chronic or acute liver failure, age greater than 80yrs.
* Patients who are unable to walk and are wheelchair bound or need assistance to walk for reasons other than CHF.
* Patients with muscular dystrophies and myopathies.
* Patients with untreated hyper or hypothyroidism.
* Patients on Dialysis.
* Patients with recent (<12 weeks) revascularization.
* Patients with recent (<12 weeks) myocardial infarction.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are scheduled for a CRT-D device
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2006-01; Primary Completion 2008-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Shift of the muscle transcriptome away from Apoptosis/Inflammation. Reversal of active apoptosis in skeletal muscle.Quality of life assessment(Minn.HF Ques) Exercise capacity (6 min walk). | 6 months

SECONDARY OUTCOMES:
Improved LV synchrony as determined by TDI, Decrease in blood markers of inflammation and Oxidative stress and catabolism. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Hranitzky, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States